CLINICAL TRIAL: NCT06921460
Title: Long-Term Protection of Vi Antibodies Induced by Vi-DT Conjugate Vaccines (Bio TCV) in Indonesian Population Compared to PQed TCV
Brief Title: Long-Term Protection of Vi Antibodies Induced by Bio TCV in Indonesian Population Compared to PQed TCV
Status: Not yet recruiting | Type: Observational
Sponsor: PT Bio Farma (Industry)
Responsible Party: Sponsor
Other Study IDs: Typhoid-0424
Record Dates: First submitted 2024-11-06; First posted 2025-04-10 (Actual); Last update posted 2025-06-03 (Actual); Status verified 2025-06

CONDITIONS: Antibody Typhoid Vaccine

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Biospecimen Retention: Samples Without DNA — Blood samples.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Test: Bio-TCV group : Blood collection for long-term protection
- Comparator: Typbar group : Blood collection for long-term protection

SUMMARY:
Typhoid fever is a serious systemic infection caused by the enteric pathogen Salmonella enterica serovar typhi. S typhi is spread by the fecal-oral route. Although largely an endemic disease, S. typhi has epidemic potential. This research aims to determine the long-term immune response after administration of one dose of Bio TCV and PQed TCV vaccines in the population in Indonesia. Research participants will be taken from research participants who complete the Bio TCV (Typhoid 0319) Phase III clinical trial research included in the Main Study Group I.

DETAILED DESCRIPTION:
Typhoid fever is a serious systemic infection caused by the enteric pathogen Salmonella enterica serovar typhi. S typhi is spread by the fecal-oral route. Although largely an endemic disease, S. typhi has epidemic potential. Data mainly from Asia, Africa and Latin America show that typhoid fever continues to be a public health problem in many developing countries, with school-age children (aged 5-15 years) disproportionately affected. In some endemic areas, children aged < 5 years show incidence rates similar to, or exceeding those, of school age children. WHO conservatively estimates the annual global incidence of typhoid fever at 21 million cases, of which 1-4% ends fatally. An estimated 90% of these deaths occur in Asia. Increasing multidrug resistance of S. typhi reduces the effective treatment options, increases treatment costs and results in higher rates of serious complications and deaths.

This research aims to determine the long-term immune response after administration of one dose of Bio TCV and PQed TCV vaccines in the population in Indonesia. Research participants will be taken from research participants who complete the Bio TCV (Typhoid 0319) Phase III clinical trial research included in the Main Study Group I. During the research, participants will make one (1) research visit to the health center for examination and blood sampling. After 5 years of being given the Typhoid vaccine, participants will be contacted by telephone to be given information about the research that will be conducted on you/your child. The research team will ask questions about the willingness to participate in the research. If they agree, a visit will be scheduled to the research site. This research is conducted by the Department of Pediatrics, Cipto Mangunkusumo Hospital, Jakarta, Dr. Soetomo Hospital, Surabaya and PT Bio Farma.

ELIGIBILITY:
Inclusion Criteria:

* Healthy
* Subject/Parents/legal guardian(s) have been informed properly regarding the study and signed the informed consent form/and informed assent form.
* Subject/parents/legal guardian(s) will commit to comply with the instructions of the investigator and the schedule of the trial.

Exclusion Criteria:

* History of uncontrolled coagulopathy or blood disorders contraindicating for phlebotomy.

Ages: 6 Months to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Subjects who previously enrolled in Phase 3 study Typhoid 0319 in Main Study I
Sampling Method: Probability Sample
Enrollment: 624 (Estimated)
Dates: Start 2025-06-15 (Estimated); Primary Completion 2025-08-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
To evaluate antibody persistence 5 years after vaccination with one dose of Vi-DT vaccine (Bio TCV), compared to PQed TCV (Typbar) | 5 years since got vaccination

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Child Health Dr. Soetomo Hospital/School of Medicine, Airlangga University, Surabaya, East Java, Jakarta, DKI Jakarta, Indonesia

IPD SHARING:
Plan to Share IPD: No